CLINICAL TRIAL: NCT01424423
Title: A Randomized, Single-blind (Investigator and Subject), Placebo-controlled, Single Ascending Dose Study Exploring the Preliminary Safety, Tolerability, and Pharmacokinetics of GSK1223249 Administered by Intravenous (IV) Infusion to Subjects With Relapsing Forms of Multiple Sclerosis, Not on Disease Modifying Therapy
Brief Title: NOGO-A in Multiple Sclerosis FTIH
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 112988
Record Dates: First submitted 2011-06-09; First posted 2011-08-29 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Multiple Sclerosis
Keywords: Safety; GSK1223249; Pharmacokinetics; Single dose escalation; anti-GSK1223249 antibodies; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — ozanezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (10):
- Subjects receiving GSK1223249 in cohort 1 (Experimental): Eligible subjects will receive intravenous infusion of GSK1223249 with a starting dose of 0.02 milligrams per kilograms, followed by 0.2, 2, 10 and 30 milligrams per kilograms, administered by a programmable syringe pump.
  Interventions: Drug: GSK1223249
- Subjects receiving placebo in cohort 1 (Placebo Comparator): Eligible subjects will receive intravenous infusion of placebo, administered by a programmable syringe pump.
  Interventions: Drug: Placebo
- Subjects receiving GSK1223249 in cohort 2 (Experimental): Eligible subjects will receive intravenous infusion of GSK1223249 with a dose of 0.2 milligrams per kilograms administered by a programmable syringe pump.
  Interventions: Drug: GSK1223249
- Subjects receiving placebo in cohort 2 (Placebo Comparator): Eligible subjects will receive intravenous infusion of placebo, administered by a programmable syringe pump.
  Interventions: Drug: Placebo
- Subjects receiving GSK1223249 in cohort 3 (Experimental): Eligible subjects will receive intravenous infusion of GSK1223249 with a dose of 2 milligrams per kilograms administered by a programmable syringe pump.
  Interventions: Drug: GSK1223249
- Subjects receiving placebo in cohort 3 (Placebo Comparator): Eligible subjects will receive intravenous infusion of placebo, administered by a programmable syringe pump.
  Interventions: Drug: Placebo
- Subjects receiving GSK1223249 in cohort 4 (Experimental): Eligible subjects will receive intravenous infusion of GSK1223249 with a dose of 10 milligrams per kilograms administered by a programmable syringe pump.
  Interventions: Drug: GSK1223249
- Subjects receiving placebo in cohort 4 (Placebo Comparator): Eligible subjects will receive intravenous infusion of placebo, administered by a programmable syringe pump.
  Interventions: Drug: Placebo
- Subjects receiving GSK1223249 in cohort 5 (Experimental): Eligible subjects will receive intravenous infusion of GSK1223249 with a dose of 30 milligrams per kilograms administered by a programmable syringe pump.
  Interventions: Drug: GSK1223249
- Subjects receiving placebo in cohort 5 (Placebo Comparator): Eligible subjects will receive intravenous infusion of placebo, administered by a programmable syringe pump.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Subjects receiving placebo in cohort 1; Subjects receiving placebo in cohort 2; Subjects receiving placebo in cohort 3; Subjects receiving placebo in cohort 4; Subjects receiving placebo in cohort 5
Drug: GSK1223249 — I.V. Infusion
  Arms: Subjects receiving GSK1223249 in cohort 1; Subjects receiving GSK1223249 in cohort 2; Subjects receiving GSK1223249 in cohort 3; Subjects receiving GSK1223249 in cohort 4; Subjects receiving GSK1223249 in cohort 5

SUMMARY:
The drug being tested in this study is GSK1223249. The drug works by inhibiting a protein that prevents nerve growth.

The trial is expected to involve approximately 36 patients. The study objective is to investigate the tolerability, safety and the way the body handles GSK1223249 after a range of single doses in patients with Multiple Sclerosis (MS).

DETAILED DESCRIPTION:
This is a phase I study of GSK1223249. The study design is randomized, placebo-controlled, double-blind, sequential dose escalation, single dose administration. Approximately 36 patients with relapsing forms of Multiple Sclerosis (having had at least two relapses over the previous 24 months, OR at least one relapse within the last 12 months, OR having had at least one documented gadolinium-enhancing lesion on brain magnetic resonance imaging (MRI) within 12 months prior to Screening) will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Suitable as determined by the Principal Investigator, based on his/her overall evaluation. A patient with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Diagnosed with a relapsing form of MS defined as either
* Relapsing Remitting MS according to revised McDonald Criteria [McDonald, 2001; Polman, 2005] plus any one of the following:

Occurrence of at least one relapse in the previous 12 months OR at least 2 relapses in the previous 24 months OR at least one documented Gd-enhancing lesion by magnetic resonance imaging (MRI) within 12 months prior to screening.

OR

-Secondary Progressive MS, plus any one of the following: Occurrence of at least one relapse in the previous 12 months OR at least 2 relapses in the previous 24 months OR at least one documented Gd-enhancing lesion by magnetic resonance imaging (MRI) within 12 months prior to screening.

* Expanded Disability Status Scale (EDSS) score ≤5.5
* Male or female between 18 and 55 years of age inclusive, at the time of signing the informed consent.

Exclusion Criteria:

* Abnormal baseline blood tests
* Treatment with interferon-beta-1b (Betaferon), interferon-beta-1a (Rebif or Avonex), or glatiramer acetate (Copaxone) within 90 days of dosing.
* Treatment with methylprednisolone or any other systemic steroids within 60 days of dosing.
* Treatment within the past 12 months or currently with any of the following agents: cyclosporine, azathioprine, methotrexate, cladribine, natalizumab (Tysabri®) or other monoclonal antibodies, murine protein, T-cell vaccination, plasmapheresis, IVI gG, ,stem cell transplantation.
* History of intolerance to acetominophen, ibuprofen, naproxen or any other non-steroidal anti-inflammatory agent which would preclude use of at least one of these during the study.
* Previous history of anaphylaxis, severe allergic reaction, or hypersensitivity to albumin or a protein-based therapeutic, including natalizumab (Tysabri) or any other monoclonal antibody. History of hypersensitivity to any of the components of the formulation.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result.
* Patients with evidence of dementia or psychiatric illness which, in the Investigator's opinion, is likely to prevent them from a full understanding of and/or compliance with the study requirements and procedures.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2010-02-11 (Actual); Primary Completion 2010-08-26 (Actual); Study Completion 2010-08-26 (Actual)

PRIMARY OUTCOMES:
The preliminary safety and tolerability of single doses of GSK1223249 | screening, baseline (pre-dose) and up to 84 days post dose
  changes in Vital signs, Electocardiogram, safety laboratory samples, adverse event (AE), neurological examination and MS relapses

SECONDARY OUTCOMES:
Single dose pharmacokinetics. | screening, baseline (pre-dose) and up to 84 days post dose
  (AUC(0-∞)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Heidelberg, Victoria, Australia

REFERENCES:
- See also: Results for study 112988 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/112988?search=study&study_ids=112988#rs